CLINICAL TRIAL: NCT01983995
Title: Prospective Pilot Study Evaluating the Inter-relationships Between Sleep Disturbance, Fatigue, Pain, and Daytime Activity in Breast Cancer Patients Starting Aromatase Inhibitor Therapy
Brief Title: Examining the Relationships Between Sleep, Fatigue, and Pain in Aromatase Inhibitor-treated Patients
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, N. Lynn Henry, Assistant Professor of Internal Medicine, Medical School, University of Michigan
Other Study IDs: HUM00078882; UMCC 2013.098 (Other: University of Michigan Cancer Center)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Aromatase Inhibitors; Actigraphy; Pain; Fatigue; Sleep quality
MeSH Terms: conditions — Breast Neoplasms; Pain; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Actigraphy: Postmenopausal women starting aromatase inhibitor therapy will undergo assessment with questionnaires and actigraphy before starting AI therapy and after 3 months of treatment.

SUMMARY:
Aromatase inhibitors are commonly prescribed for treatment of postmenopausal women with breast cancer. These medications can cause side effects in some women, and occasionally they can be quite bothersome. We are doing a study to better understand the side effects of aromatase inhibitors so that we can hopefully treat them better or possibly prevent them. In particular, we are interested in pain and difficulty sleeping. This study is designed to assess the effect of aromatase inhibitors on pain, sleep quality, and fatigue and the interplay of these side effects and their subsequent impact on daily activity. Each participant will fill out a series of questionnaires about pain, sleep quality, and fatigue and will also complete a sleep diary and wear an actigraphy watch for 10 days before starting an aromatase inhibitor and after taking it for 3 months. We hope to learn more about these symptoms so we can better manage medication toxicity in the future.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 50 years or older, postmenopausal.
* Patients with histologically proven stage 0-III invasive carcinoma of the breast that is estrogen receptor and/or progesterone receptor positive by immunohistochemical staining, who are planning to start treatment with a standard dose of aromatase inhibitor (AI) therapy.
* Subjects must have undergone surgical resection of their primary tumor, as indicated. The most recent surgery must have been performed at least 4 weeks before the baseline evaluation and no additional surgeries (including reconstructive procedures) should be planned during study participation.
* Cytoxic chemotherapy, if applicable, must have been completed at least 4 weeks before the baseline evaluation.
* Radiation therapy, if applicable, must have been completed at least 2 weeks before baseline evaluation.
* Eastern Cooperative Oncology Group performance status 0-2.
* Ability to operate the accelerometer

Exclusion Criteria:

* Diagnosis of sleep apnea or restless leg syndrome.
* Use of a wheelchair for ambulation most of the time.
* Second or third shift workers or other non-traditional sleep schedules.
* History of medical arthritic disease that could confound or interfere with evaluation of pain or activity level, including but not limited to inflammatory arthritis (rheumatoid arthritis, systemic lupus, spondyloarthropathy, psoriatic arthritis, polymyalgia rheumatica), Parkinson's disease, and cancer involving the bone.
* Serious or unstable medical condition that could likely lead to hospitalization during the course of the study or compromise study participation

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Michigan Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting an actigraphy study with breast cancer patients | 3 months
  Feasibility will be measured by the proportion of breast cancer patients who are starting aromatase inhibitor therapy who complete baseline and 3 month assessment questionnaires and also enter actigraphy data correctly at least 85% of the time.

SECONDARY OUTCOMES:
Association between patient-reported sleep quality, fatigue, and pain and objective actigraphy measurements. | 3 months
  We will evaluate patterns of symptoms reported by subjects and the apparent impact of these symptoms on both daytime function and sleep quality.
Change in pain, fatigue, sleep disturbance, and daytime activity with 3 months of aromatase inhibitor therapy | 3 Months
  We will analyze the change in sleep, pain, fatigue, and symptom severity index between baseline and 12 weeks. We will correlate changes in symptoms from baseline to 12 weeks with actigraphy activity.

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States